CLINICAL TRIAL: NCT01557335
Title: A Randomized, Open-Label, Cross-Over, Study to Evaluate the Inhibitory Effect of Clopidogrel, EC Aspirin 81 mg and EC Omeprazole 40 mg All Dosed Concomitantly and PA32540 and Clopidogrel Dosed Separately on Platelet Aggregation in Healthy Volunteers
Brief Title: A Study to Evaluate Platlet Aggregation of Clopidogrel, EC Aspirin 81 mg, EC Omeprazole 40 mg Compare to PA32540
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: POZEN (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PA32540-111
Record Dates: First submitted 2012-03-13; First posted 2012-03-19 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Platelet Aggregation
Keywords: To evaluate adenosine diphosphate (ADP)-induced platelet aggregation
MeSH Terms: interventions — Clopidogrel; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel (Plavix®) and PA32540 (Experimental): PA32540 and Clopidogrel (Plavix®) tablet, 10 hours post PA32540
  Interventions: Drug: Plavix® and PA32540
- EC aspirin, EC omeprazole, Clopidogrel (Active Comparator)
  Interventions: Drug: EC aspirin (Bayer®) ,EC omeprazole (Prilosec®) , Clopidogrel (Plavix®)

INTERVENTIONS:
Drug: Plavix® and PA32540 — one Plavix® 300 mg loading dose in the PM of Day 1 one Plavix® 75 mg maintenance dose in the PM of Days 2-7 PA32540(delayed release aspirin 325 mg plus immediate release omeprazole 40 mg)
  Arms: Clopidogrel (Plavix®) and PA32540
Drug: EC aspirin (Bayer®) ,EC omeprazole (Prilosec®) , Clopidogrel (Plavix®) — One EC aspirin (Bayer®) 81 mg tablet plus one EC omeprazole (Prilosec®) 40 mg capsule plus one Clopidogrel (Plavix®) tablet of 300 mg (loading dose) all One EC aspirin (Bayer®) 81 mg tablet plus one EC omeprazole (Prilosec®) 40 mg capsule plus one Clopidogrel (Plavix®) tablet of 75 mg (maintenance dose) all taken concomitantly in the AM of Days 2-7
  Arms: EC aspirin, EC omeprazole, Clopidogrel

SUMMARY:
This study is designed to provide data on platelet aggregation of PA32540 plus clopidogrel dosed separately compared to EC aspirin 81 mg plus EC omeprazole 40 mg plus clopidogrel dosed concomitantly.

DETAILED DESCRIPTION:
PA32540 is proposed for the secondary prevention of cardio- and cerebrovascular events in patients at risk for developing aspirin-associated gastric ulcers.

Aspirin 81 mg taken concomitantly with clopidogrel 75 mg as maintenance doses is standard of care in some patients with cardiovascular disease. The combination of aspirin and clopidogrel, however, significantly increases the risk for bleeding events. To mitigate upper gastrointestinal bleeding events, these patients would require the use of a proton pump inhibitor. For that reason, the reference arm in this study uses Prilosec® 40 mg as a comparator - the same proton pump inhibitor at the same dose level.

The primary objective is to evaluate adenosine diphosphate (ADP)-induced platelet aggregation following administration of clopidogrel, EC aspirin 81 mg and EC omeprazole 40 mg, all dosed concomitantly, and PA32540 and clopidogrel dosed separately

ELIGIBILITY:
Inclusion Criteria:

* Male or non-lactating, non-pregnant female subjects who are 40 years or older at the time of initial dosing

  --Physical status within normal limits for age and consistent with observations at Screening
* Able to understand and comply with study procedures required and able and willing to provide written informed consent prior to any study procedures being performed

Exclusion Criteria:

* History of hypersensitivity, allergy or intolerance to omeprazole or other proton-pump inhibitors (PPIs)
* History of hypersensitivity, allergy or intolerance to aspirin or any NSAID and/or a history of NSAID-induced symptoms of asthma, rhinitis, and/or nasal polyps
* History of hypersensitivity or intolerance to clopidogrel
* History of hepatitis B or C, a positive test for hepatitis B surface antigen, hepatitis C antibody, a history of human immunodeficiency virus (HIV) infection or demonstration of HIV antibodies
* History of malignancy, treated or untreated, within the past five years, with the exception of successfully treated basal cell or squamous cell carcinoma of -Evidence of uncontrolled, or unstable cardio- or cerebrovascular disorder, which in the Investigator's opinion, would endanger a subject if he/she were to participate in the study
* Presence of an uncontrolled acute, or a chronic medical illness, e.g., GI disorder, diabetes, hypertension, thyroid disorder, bleeding disorder, infection, which in the Investigator's opinion would endanger a subject if he/she were to participate in the study or interfere with the objective of this study
* Schizophrenia or bipolar disorder
* GI disorder or surgery leading to impaired drug absorption
* < 70% platelet aggregation at Screening
* Donation of blood or plasma within 4 weeks of the study
* PPI use or any enzyme inducing/inhibiting agents within 4 weeks prior to dosing
* Taking any antiplatelet drug within 2 weeks of the screening visit or during the study, or more than two 325 mg doses of aspirin or more than 2 doses of any other NSAIDs within 14 days prior to the screening visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Evaluate adenosine diphosphate (ADP)-induced platelet aggregation | 7 days
  To evaluate adenosine diphosphate (ADP)-induced platelet aggregation following administration of clopidogrel, EC aspirin 81 mg and EC omeprazole 40 mg, all dosed concomitantly, and PA32540 and clopidogrel dosed separately.
  The endpoint measure is IPA (Individual Platelet Aggregation)at day 7 and PA0 is the platelet aggregation at baseline. The IPA will be analyzed using analyses of variance (ANOVA).

SECONDARY OUTCOMES:
Evaluate arachidonic acid (AA)-induced platelet aggregation | 7 days
  To evaluate arachidonic acid (AA)-induced platelet aggregation following administration of clopidogrel, EC aspirin 81 mg and EC omeprazole 40 mg, all dosed concomitantly, and PA32540 and clopidogrel dosed separately.
  The secondary endpoint is the IPA (Individual Platelet Aggregation) and will be analyzed using the same methodology as the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Zimmerman, Study Director — POZEN
Locations (1):
- Sinai Center for Thrombosis Research, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Gurbel PA, Bliden KP, Fort JG, Jeong YH, Shuldiner A, Chai S, Gesheff T, Antonino M, Gesheff M, Zhang Y, Tantry US. Spaced administration of PA32540 and clopidogrel results in greater platelet inhibition than synchronous administration of enteric-coated aspirin and enteric-coated omeprazole and clopidogrel. Am Heart J. 2013 Feb;165(2):176-82. doi: 10.1016/j.ahj.2012.07.032. Epub 2012 Dec 4. PMID 23351820